CLINICAL TRIAL: NCT02268305
Title: The Use of Methylsulfonylmethane (MSM) in the Treatment of Low Back Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20140075H
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — dimethyl sulfone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSM 1000mg twice a day (6000 mgs) (Experimental): Group 1 will take by mouth three 1000 mg capsules twice a day (6000 mgs) of MSM plus standard of care naproxen
  Interventions: Drug: MSM 1000mg twice a day (6000 mgs)
- Placebo capsules twice a day (Placebo Comparator): Group 2 will take by mouth three placebo capsules twice a day plus standard of care naproxen
  Interventions: Other: Placebo capsules twice a day

INTERVENTIONS:
Drug: MSM 1000mg twice a day (6000 mgs) — MSM is believed to have anti-inflammatory properties. MSM is a largely tasteless, odorless, white, crystalline solid which is water soluble. It occurs naturally in the environment and is synthesized in the human body as a byproduct of dietary DMSO.
  Other Names: Methylsulfonylmethane
  Arms: MSM 1000mg twice a day (6000 mgs)
Other: Placebo capsules twice a day — Placebo is a capsule filled with rice flour.
  Other Names: Placebo
  Arms: Placebo capsules twice a day

SUMMARY:
The investigators are studying whether MSM plus standard of care naproxen improves symptoms of lower back pain compared to standard of care naproxen plus placebo. Subjects will be randomized into 1 of 2 groups. Group 1 will take by mouth 6000 milligrams (mgs) of MSM plus standard of care naproxen. Group 2 will take by mouth placebo capsules plus standard of care naproxen. Subjects will be instructed to take their study pills for 12 weeks and record on a study diary. They will then be followed up for one final visit 4 weeks later. RMDQ, PIQ-6, pain level, comprehensive metabolic panel (CMP), complete blood count (CBC) will be assessed at 4 week intervals for 12 weeks. Subjects' participation will last 16 weeks.

DETAILED DESCRIPTION:
We will recruit male and female MOFMC DoD beneficiaries between the ages of 18-65 years old with symptoms of lower back pain from any of the clinics at the MOFMC at Nellis Air Force Base. Patients taking Muscle relaxers of any type, Non-steroidal anti-inflammatory agents (NSAIDs), Tramadol, Gabapentin, Pregabalin, agree to wash out for two weeks prior to entering the study.

Screening Visit:

* Obtain signed Informed Consent Document and HIPAA Authorization.
* Review inclusion/exclusion criteria.
* Record: name, race ethnicity, race, date of birth, age, sex, height (in inches), weight (in pounds), blood pressure, email address, phone number, history of lower back surgeries, medical history, concomitant medications, and record the amount of naproxen prescribed as standard of care.
* Subjects will have the following research-driven blood test drawn via 1 venipuncture (5-10 mls, approximately 1-2 teaspoons of blood drawn for each test) which include:

  * Women of childbearing potential will have a serum pregnancy test.
  * Comprehensive metabolic panel (liver function, renal function, plasma glucose tests).

    *Subjects who have had a comprehensive metabolic panel test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.
  * Complete Blood Count. *Subjects who have had a complete blood count test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.

Visit 1/Day 1 (within 1 week of Screening Visit):

* Subjects will be randomized by the research coordinator. We will use a minimization/dynamic determination randomization (see attached explanation of minimization/dynamic determination) technique to ensure roughly equal sample sizes. Both subjects and investigators will be blinded to the study group assignments:

  * Group 1 will take by mouth three 1000 mg capsules twice a day (6000 mgs) of MSM plus standard of care naproxen.
  * Group 2 will take by mouth three placebo capsules twice a day plus standard of care naproxen.
* Subjects will be asked to complete the following questionnaires:

  * RMDQ
  * PIQ-6
* Subjects will be asked "On a scale of 0-10, with 10 being the worst pain, what is your current level of pain".
* Subjects will be given a 12 week supply of the study pills and reminded to take the pills as instructed.
* Subjects will be given a Study Diary and will be instructed to record any missed dose of their study pills, record how much standard of care naproxen taken, and to bring the Study Diary to next visit.

Visit 2/Week 4:

* Record: Weight (in pounds), blood pressure, history of lower back surgeries, medical history, and concomitant medications.
* Subjects will be asked to complete the following questionnaires:

  * RMDQ
  * PIQ-6
* Subjects will be asked "On a scale of 0-10, with 10 being the worst pain, what is your current level of pain".
* Research staff will record whether subject had any side effects to report.
* Research staff will collect the subject's Study Diary, issue them a new one, and remind them to bring it with them to the next study visit.
* Research staff will remind subjects to take the pills as instructed.
* Subjects will have the following research-driven blood test drawn via 1 venipuncture (5-10 mls, approximately 1-2 teaspoons of blood drawn for each test) which include:

  * Comprehensive metabolic panel (liver function, renal function, plasma glucose tests).

    *Subjects who have had a comprehensive metabolic panel test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.
  * Complete Blood Count.

    * Subjects who have had a complete blood count test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.

Visit 3/Week 8:

* Record: Weight (in pounds), blood pressure, history of lower back surgeries, medical history, and concomitant medications.
* Subjects will be asked to complete the following questionnaires:

  * RMDQ
  * PIQ-6
* Subjects will be asked "On a scale of 0-10, with 10 being the worst pain, what is your current level of pain".
* Research staff will record whether subject had any side effects to report.
* Research staff will collect the subject's Study Diary, issue them a new one, and remind them to bring it with them to the next study visit.
* Research staff will remind subjects to take the pills as instructed and to return the bottle to the research staff at the next visit.
* Subjects will have the following research-driven blood test drawn via 1 venipuncture (5-10 mls, approximately 1-2 teaspoons of blood drawn for each test) which include:

  * Comprehensive metabolic panel (liver function, renal function, plasma glucose tests).

    *Subjects who have had a comprehensive metabolic panel test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.
  * Complete Blood Count. *Subjects who have had a complete blood count test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.

Visit 4/Week 12 *SUBJECTS STOP TAKING STUDY PILLS AT THIS VISIT:

* Record: Weight (in pounds), blood pressure, history of lower back surgeries, medical history, and concomitant medications.
* Subjects will be asked to complete the following questionnaires:

  * RMDQ
  * PIQ-6
* Subjects will be asked "On a scale of 0-10, with 10 being the worst pain, what is your current level of pain".
* Research staff will record whether subject had any side effects to report.
* Research staff will collect the subject's Study Diary.
* Research staff will collect the study pills.
* Subjects will have the following research-driven blood test drawn via 1 venipuncture (5-10 mls, approximately 1-2 teaspoons of blood drawn for each test) which include:

  * Comprehensive metabolic panel (liver function, renal function, plasma glucose tests).

    *Subjects who have had a comprehensive metabolic panel test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.
  * Complete Blood Count. *Subjects who have had a complete blood count test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.

Final Visit 5/Week 16:

* Record: Weight (in pounds), blood pressure, history of lower back surgeries, medical history, and concomitant medications.
* Subjects will be asked to complete the following questionnaires:

  * RMDQ
  * PIQ-6
* Subjects will be asked "On a scale of 0-10, with 10 being the worst pain, what is your current level of pain".
* Research staff will record whether subject had any side effects to report.
* Subjects will have the following research-driven blood test drawn via 1 venipuncture (5-10 mls, approximately 1-2 teaspoons of blood drawn for each test) which include:

  * Comprehensive metabolic panel (liver function, renal function, plasma glucose tests).

    *Subjects who have had a comprehensive metabolic panel test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.
  * Complete Blood Count. *Subjects who have had a complete blood count test within the one week prior to this visit will not need to have this test repeated unless they are abnormal.

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion:

DoD beneficiaries between the ages of 18-65 years old Symptoms of Low Back Pain greater than 12 weeks duration Patients with a history of lower back surgery may be included

Exclusion:

DoD beneficiaries less than 18 years old or greater than 65 years old

Lower back pain caused by any of the following:

Infection Tumor Osteoporosis Ankylosing spondylitis Fracture Deformity Inflammatory process Cauda equina syndrome Treated or untreated central nervous system impairment

Meeting the criteria for surgery, including:

progressive motor deficit sphincter impairment from neurological cause disabling sciatic pain (in the absence of backache) lasting 6 weeks or more that is attributed to a compromised nerve root and demonstrated by magnetic resonance imaging or computed tomography Oncologic disease during the previous 5 years Unexplained weight loss, fever, or chills Diagnosed upper urinary tract infection within last 28 days Patients identified during standard of care interview to have a history of intravenous drug use.

Immunocompromised host

A severe comorbidity to include:

determining overall well-being (e.g. painful disabling arthritic hip joints) Cirrhosis Ongoing dialysis Radiating symptoms to lower extremities (sciatica) History of bleeding disorders History of high blood pressure History of heart, kidney, liver or ulcer disease Allergic to analgesics or Non-steroidal anti inflammatory agents (NSAIDs) Pregnant or breastfeeding Initial pain rating of greater than 8/10 on initial intake evaluation If any of the components of the comprehensive metabolic panel are outside the Nellis clinical laboratory reference ranges, the subject will be excluded from the study

If any of these four components of the complete blood count are outside of the Nellis clinical laboratory reference ranges, the subject will be excluded from the study:

White blood cell count Hemoglobin Hematocrit Platelets

Patients taking any of the following medications are excluded from participating, unless they agree to wash out for two weeks prior to entering the study:

Muscle relaxers of any type Non-steroidal anti-inflammatory agents (NSAIDs) * Patients taking naproxen must agree to wash out for two weeks prior to entering the study, but can begin taking it again, as prescribed, after Visit 1 where a baseline pain assessment is performed.

Tramadol Gabapentin Pregabalin Glucosamine Narcotic pain medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, MD, Principal Investigator — Mike O'Callaghan Federal Medical Center
Locations (1):
- Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 86 subjects analyzed.
Period: Overall Study
Arm/Group | MSM 1000mg Twice a Day (6000 Mgs) | Placebo Capsules Twice a Day
Started | 50 | 50
Completed | 46 | 40
Not Completed | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSM 1000mg Twice a Day (6000 Mgs) | Placebo Capsules Twice a Day | Total
Number analyzed (Participants) | 46 | 40 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 40 | 86
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 30 | 29 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 6 | 15
  White | 21 | 25 | 46
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 46 | 40 | 86

OUTCOME MEASURES:

1. Primary Outcome: Pain Level
Description: decrease in pain via analogue pain scale of 0-10 (with 10 being the worst pain)
Time Frame: 16 weeks (Weeks 0, 4, 8, 12, and 16)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MSM 1000mg Twice a Day (6000 Mgs) | Placebo Capsules Twice a Day
Number analyzed (Participants) | 46 | 40
score on a scale
  Visual Analogue Scale Week 0 | 3.4 (1.5) | 3.7 (2.0)
  Visual Analogue Scale Week 4 | 2.8 (1.5) | 2.9 (2.5)
  Visual Analogue Scale Week 8 | 3.0 (1.6) | 3.1 (2.4)
  Visual Analogue Scale Week 12 | 2.7 (1.4) | 3.2 (2.4)
  Visual Analogue Scale Week 16 | 3.0 (1.7) | 3.4 (2.4)

2. Secondary Outcome: Roland-Morris Disability Questionnaire
Description: symptoms of lower back pain. 0 (no disability) to 24 (max. disability).
Time Frame: 16 weeks (Weeks 0, 4, 8, 12, and 16)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MSM 1000mg Twice a Day (6000 Mgs) | Placebo Capsules Twice a Day
Number analyzed (Participants) | 46 | 40
score on a scale
  Roland Morris Disability Questionnaire Week 0 | 8.0 (4.2) | 8.4 (5.1)
  Roland Morris Disability Questionnaire Week 4 | 5.8 (4.3) | 6.9 (5.8)
  Roland Morris Disability Questionnaire Week 8 | 5.5 (3.9) | 6.7 (5.5)
  Roland Morris Disability Questionnaire Week 12 | 5.4 (4.2) | 6.9 (4.2)
  Roland Morris Disability Questionnaire Week 16 | 5.9 (4.4) | 6.8 (5.7)

3. Secondary Outcome: Pain Impact Questionnaire-6
Description: 6-item questionnaire measuring pain's interference with life activities. The total possible score of the PIQ-6 ranges from 40-78 points, where lower scores indicate less pain interference.
Time Frame: 16 weeks (Weeks 0, 4, 8, 12, and 16)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MSM 1000mg Twice a Day (6000 Mgs) | Placebo Capsules Twice a Day
Number analyzed (Participants) | 46 | 40
score on a scale
  Pain Impact Questionnaire Week 0 | 60.8 (5.0) | 60.2 (6.9)
  Pain Impact Questionnaire Week 4 | 56.4 (6.5) | 56.7 (8.5)
  Pain Impact Questionnaire Week 8 | 56.0 (6.4) | 57.2 (9.6)
  Pain Impact Questionnaire Week 12 | 56.5 (6.4) | 56.3 (9.3)
  Pain Impact Questionnaire Week 16 | 57.0 (6.9) | 57.8 (8.6)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | MSM 1000mg Twice a Day (6000 Mgs) | Placebo Capsules Twice a Day
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 2/50 | 2/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSM 1000mg Twice a Day (6000 Mgs) (N=50) | Placebo Capsules Twice a Day (N=50)
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT02268305/Prot_SAP_000.pdf